CLINICAL TRIAL: NCT01251757
Title: Promoting Adherence to Improve Effectiveness of Cardiovascular Disease Therapies (PATIENT)
Brief Title: Promoting Adherence to Improve Effectiveness of Cardiovascular Disease Therapies
Acronym: PATIENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Kaiser Foundation Hospitals, Center for Health Research (Other); Johns Hopkins University (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01HS019341-01 (AHRQ)
Record Dates: First submitted 2010-11-30; First posted 2010-12-02 (Estimated); Results first posted 2017-02-01 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Mellitus; Cardiovascular Disease
Keywords: diabetes; cardiovascular disease; randomized clinical trial; medication adherence; health information technology; adult; telephone calls; IVR
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Usual Care (UC) (No Intervention): Participants in this arm received their usual care with no restrictions.
- Interactive Voice Recognition (IVR) (Active Comparator): automated phone calls
  Interventions: Other: Interactive Voice Recognition (IVR) phone calls
- Enhanced IVR (IVR+) (Active Comparator): automated phone calls & Educational mailings and follow-up for nonadherence
  Interventions: Other: Interactive Voice Recognition (IVR) phone calls; Other: Educational mailings and follow-up for nonadherence

INTERVENTIONS:
Other: Interactive Voice Recognition (IVR) phone calls — The IVR intervention consisted of automated phone calls designed to educate participants about their medications and to assist them in refilling their prescriptions. The calls fell into two basic types: simple refill reminders and "tardy" calls for those who were overdue for a refill. Calls occured monthly and were triggered by dispensing information in the electronic medical record (EMR). Call features included the ability to transfer individuals to Kaiser's automated prescription refill service as well as to care managers. Although the calls were triggered by and focused on use of ACE inhibitors, ARBs and statins, they also included reminders to use aspirin, which is known to also be effective for secondary prevention in this patient population.
  Other Names: automated phone calls
  Arms: Enhanced IVR (IVR+); Interactive Voice Recognition (IVR)
Other: Educational mailings and follow-up for nonadherence — Participants received bimonthly educational materials by mail. In addition, patients received mailed refill reminder letters and their providers were notified electronically if the patients failed to refill in response to the automated calls. The educational mailings included personalized health information such as the participant's cholesterol and blood pressure readings, as well as tools for improving adherence such as frequently asked questions (FAQs) about their medications, a pocket-sized calendar for tracking refills with pertinent phone numbers and web site information and space for them to write their medical record number and prescription numbers.
  Other Names: mail follow-up for nonadherence; educational mailings
  Arms: Enhanced IVR (IVR+)

SUMMARY:
The purpose of this randomized clinical trial is to determine whether two low-intensity, technology based interventions, when compared to each other and to usual care, improve adherence to selected medications that are used to treat people with cardiovascular disease (CVD) and diabetes.

DETAILED DESCRIPTION:
The frequent failure of patients to adhere to long-term medication regimens remains the single greatest challenge for chronic-disease management. Many studies have linked medication non-adherence to treatment failure; unnecessary and dangerous intensification of therapy; and excess health care costs, hospitalizations, and deaths. Although some interventions have been shown to significantly enhance medication adherence, the strategies used are often complex, labor-intensive, and of variable effectiveness. Simple interventions designed to make small-but-significant improvements in population-based adherence may thus offer a novel, cost-effective, and easily-disseminated alternative to current approaches for enhancing adherence. The proposed PATIENT study will use health information technology (automated phone calls and access to an electronic medical record) to test two such interventions and compare them to each other and to usual care alone.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40 years or older as of time of randomization.
* Flagged in KP's databases as having either diabetes or atherosclerotic cardiovascular disease(defined as coronary artery disease, peripheral vascular disease, or a history of atherosclerotic stroke) at the time of randomization
* At least one dispensing of an ACEI, ARB, or statin from a Kaiser Permanente (KP) outpatient pharmacy during the baseline year.
* Suboptimal adherence ((MPR<0.9) to either statins or ACEI/ARBs during the baseline year
* Continuous membership in KP for the 12 months prior to randomization.
* Qualified for an intervention call at the time of randomization.

Exclusion Criteria:

* Evidence in the electronic medical record (EMR) of allergy or intolerance to statins or ACE inhibitors/ARBs
* medical conditions that would contraindicate use of statins or ACEI/ARBs
* Absence of either a phone number or mailing address in the EMR
* for Kaiser Permanente Hawaii, clinics whose patients tend to fill prescriptions primarily at non-KP pharmacies
* on Kaiser Permanente's "do not contact" list or in other research studies that could add undue burden

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21752 (Actual)
Dates: Start 2011-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William M Vollmer, PhD, Principal Investigator — Center for Health Research, Kaiser Permanente Northwest
Locations (3):
- United States (3):
  - Center for Health Research, Kaiser Permanente Southeast, Atlanta, Georgia
  - Center for Health Research, Kaiser Permanente Hawaii, Honolulu, Hawaii
  - Center for Health Research, Kaiser Permanente Northwest, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No
At the request of AHRQ we did not create a formal public data release.

REFERENCES:
- [Result] Vollmer WM, Owen-Smith AA, Tom JO, Laws R, Ditmer DG, Smith DH, Waterbury AC, Schneider JL, Yonehara CH, Williams A, Vupputuri S, Rand CS. Improving adherence to cardiovascular disease medications with information technology. Am J Manag Care. 2014 Nov;20(11 Spec No. 17):SP502-10. PMID 25811824
- [Result] Smith DH, O'Keeffe-Rosetti M, Owen-Smith AA, Rand C, Tom J, Vupputuri S, Laws R, Waterbury A, Hankerson-Dyson DD, Yonehara C, Williams A, Schneider J, Dickerson JF, Vollmer WM. Improving Adherence to Cardiovascular Therapies: An Economic Evaluation of a Randomized Pragmatic Trial. Value Health. 2016 Mar-Apr;19(2):176-84. doi: 10.1016/j.jval.2015.11.013. Epub 2016 Feb 12. PMID 27021751
- [Result] Owen-Smith AA, Smith DH, Rand CS, Tom JO, Laws R, Waterbury A, Williams A, Vollmer WM. Difference in Effectiveness of Medication Adherence Intervention by Health Literacy Level. Perm J. 2016 Summer;20(3):15-200. doi: 10.7812/TPP/15-200. Epub 2016 Jun 29. PMID 27352409

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care (UC): Participants in this arm had full access to all care they were normally entitled to as part of usual care
- Interactive Voice Recognition (IVR): In addition to their usual care, participants in the Interactive Voice Recognition (IVR) arm received automated phone calls, triggered by dispensing events in the electronic medical record (EMR), to educate patients about their medications and assist them in refilling their prescriptions.
  The calls fell into two basic types: simple refill reminders and "tardy" calls for those who were overdue for a refill. Calls occured monthly and were triggered by dispensing information in the EMR. Call features included the ability to transfer individuals to Kaiser's automated prescription refill service as well as to care managers. Although the calls were triggered by and focused on use of ACE inhibitors, ARBs and statins, they also included reminders to use aspirin, which is known to also be effective for secondary prevention in this patient population.
- Enhanced IVR (IVR+): Participants in the IVR+ arm received all components of the IVR intervention and in addition were mailed educational materials bimonthly during the intervention. In addition, both IVR+ participants and their primary care providers received mailed notifications when they did not fill their medications in response to the automated calls.
  The educational mailings included personalized health information such as the participant's cholesterol and blood pressure readings, as well as tools for improving adherence such as FAQs about their medications, a pocket-sized calendar for tracking refills with pertinent phone numbers and web site information and space for them to write their medical record number and prescription numbers.
Period: Overall Study
Arm/Group | Usual Care (UC) | Interactive Voice Recognition (IVR) | Enhanced IVR (IVR+)
Started | 7255 (Separate analyses were done for statin users and ACEI/ARB users. This is the combined N.) | 7247 (Separate analyses were done for statin users and ACEI/ARB users. This is the combined N.) | 7250 (Separate analyses were done for statin users and ACEI/ARB users. This is the combined N.)
Completed | 7255 (mean (SD) duration of follow-up was 9.7 (2.3) mos, but we computed an adherence score for everyone.) | 7247 (mean (SD) duration of follow-up was 9.6 (2.4) mos, but we computed an adherence score for everyone.) | 7250 (mean (SD) duration of follow-up was 9.6 (2.5) mos, but we computed an adherence score for everyone.)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care (UC) | Interactive Voice Recognition (IVR) | Enhanced IVR (IVR+) | Total
Number analyzed (Participants) | 7255 | 7247 | 7250 | 21752
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (12.2) | 63.6 (12.1) | 63.5 (12.2) | 63.6 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3432 | 3370 | 3415 | 10217
  Male | 3823 | 3877 | 3835 | 11535
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 51 | 43 | 44 | 138
  Asian | 1270 | 1290 | 1254 | 3814
  Native Hawaiian or Other Pacific Islander | 798 | 819 | 783 | 2400
  Black or African American | 1168 | 1094 | 1109 | 3371
  White | 3403 | 3399 | 3408 | 10210
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 565 | 602 | 652 | 1819
Region of Enrollment [Number; unit: participants]
  United States | 7255 | 7247 | 7250 | 21752
ever smokers [Number; unit: participants]
  yes | 3482 | 3537 | 3560 | 10579
  no | 3773 | 3710 | 3690 | 11173
co-morbid diabetes mellitus [Number; unit: participants]
  yes | 5666 | 5703 | 5626 | 16995
  no | 1589 | 1544 | 1624 | 4757
co-morbid cardiovascular disease [Number; unit: participants]
  yes | 2626 | 2616 | 2661 | 7903
  no | 4629 | 4631 | 4589 | 13849
target medication use [Number; unit: participants]
  statin only | 2924 | 2870 | 2922 | 8716
  ACEI/ARB only | 1770 | 1790 | 1820 | 5380
  statin and ACEI/ARB | 2561 | 2587 | 2508 | 7656

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Statins
Description: We used a modification of the Medication Possession Ratio (MPR) as our primary outcome measure. The MPR is computed as the number of days' supply of medication dispensed during a given time window divided by the time between the first dispensing in the window and the end of the window. Our modified MPR (mMPR) also accounted for medication that was on hand at the start of the window and ignored any days' supply that would extend beyond the end of the window.
  We used medication dispensing data from the Kaiser outpatient pharmacies to calculate a modified medication possession ratio (mMPR) for statins among the subset of randomized participants who were using these drugs. Nominally mMPR provides an estimate of the proportion of days during the follow-up period during which the participant was adherent to their prescribed medications.
Time Frame: 12 months post randomization
Population: All randomized participants who were taking statins at the time of randomization
Measure: Mean (Standard Deviation); unit: mMPR as a fraction
Groups:
- Usual Care (UC): statin users in UC arm
- Interactive Voice Recognition (IVR): statin users in IVR arm
- Enhanced IVR (IVR+): statin users in IVR+ arm
Arm/Group | Usual Care (UC) | Interactive Voice Recognition (IVR) | Enhanced IVR (IVR+)
Number analyzed (Participants) | 5484 | 5453 | 5429
mMPR as a fraction
  overall | 0.55 (0.35) | 0.57 (0.34) | 0.58 (0.34)
  baseline adherence <= 0.40: number analyzed (Participants) | 1880 | 1827 | 1842
  baseline adherence <= 0.40 | 0.38 (0.37) | 0.41 (0.36) | 0.41 (0.36)
  baseline adherence 0.4-0.75: number analyzed (Participants) | 3165 | 3141 | 3122
  baseline adherence 0.4-0.75 | 0.61 (0.31) | 0.63 (0.31) | 0.65 (0.30)
  baseline adherence 0.75-0.90: number analyzed (Participants) | 439 | 485 | 465
  baseline adherence 0.75-0.90 | 0.75 (0.27) | 0.77 (0.27) | 0.75 (0.29)
Statistical Analysis 1: Comparison: Usual Care (UC) vs Interactive Voice Recognition (IVR); We conducted separate primary analyses of each of IVR and IVR+ versus usual care at the .025 level of significance to assure a trial-wide error rate of .05. This analysis summary is for the IVR versus UC comparison only. Also, we only report results here for the full sample, and not also separately for the 3 baseline adherence level groups; Test type: Superiority or Other; p < .001, Regression, Linear; adjusted for site, gender, age, total number of prescription medications patient is taking, comorbid diabetes/CVD, and baseline statin adherence; Mean Difference (Final Values) = 0.022, 95% CI 2-sided [0.011 to 0.034] — Adjusted difference in adherence for IVR group versus UC group, calculated as IVR - UC
Statistical Analysis 2: Comparison: Usual Care (UC) vs Enhanced IVR (IVR+); We conducted separate primary analyses of each of IVR and IVR+ versus usual care at the .025 level of significance to assure a trial-wide error rate of .05. This analysis summary is for the IVR+ versus UC comparison only. Also, we only report results here for the full sample, and not also separately for the 3 baseline adherence level groups; Test type: Superiority or Other; p < .001, Regression, Linear; adjusted for site, gender, age, total number of prescription medications participant is taking, comorbid diabetes/CVD, and baseline statin adherence; Mean Difference (Final Values) = 0.030, 95% CI 2-sided [0.019 to 0.042] — Adjusted difference in adherence for IVR+ group versus UC group, calculated as IVR+ - UC

2. Primary Outcome: Adherence to Angiotensin-Converting Enzyme Inhibitors (ACEIs) and Angiotensin Receptor Blockers (ARBs)
Description: We used medication dispensing data from the Kaiser outpatient pharmacies to calculate a modified medication possession ratio (mMPR) for the subset of randomized participants who were using ACEIs or ARBs. Nominally mMPR provides an estimate of the proportion of days during the follow-up period during which the participant was adherent to their prescribed medications.
Time Frame: 12 months post randomization
Population: All randomized participants who were taking an ACEI or an ARB at the time of randomization
Measure: Mean (Standard Deviation); unit: mMPR expressed as a fraction
Groups:
- Usual Care (UC): ACEI/ARB users in UC arm
- Interactive Voice Recognition (IVR): ACEI/ARB users in IVR arm
- Enhanced IVR (IVR+): ACEI/ARB users in IVR+ arm
Arm/Group | Usual Care (UC) | Interactive Voice Recognition (IVR) | Enhanced IVR (IVR+)
Number analyzed (Participants) | 4330 | 4370 | 4323
mMPR expressed as a fraction
  overall | 0.57 (0.36) | 0.59 (0.35) | 0.61 (0.34)
  baseline adherence <=0.50 | 0.45 (0.37) | 0.47 (0.37) | 0.50 (0.36)
  baseline adherence 0.50-0.75 | 0.69 (0.30) | 0.70 (0.29) | 0.71 (0.29)
  baseline adherence 0.75-0.90 | 0.76 (0.26) | 0.76 (0.28) | 0.77 (0.29)
Statistical Analysis 1: Comparison: Usual Care (UC) vs Interactive Voice Recognition (IVR); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.022, Regression, Linear; Adjusted for site, gender, age, total number of prescription medications participant was taking, comorbid diabetes/CVD, baseline ACEI/ARB adherence; Mean Difference (Final Values) = 0.016, 95% CI 2-sided [0.002 to 0.029] — Adjusted difference in adherence for IVR+ group versus UC group, calculated as IVR+ - UC
Statistical Analysis 2: Comparison: Usual Care (UC) vs Enhanced IVR (IVR+); [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < .001, Regression, Linear; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.037, 95% CI 2-sided [0.023 to 0.050] — Adjusted difference in adherence for IVR+ group versus UC group, calculated as IVR+ - UC

3. Secondary Outcome: Percentage With Good (>80%) Statin Adherence
Description: Binary indicator of good statin adherence, defined as an mMPR>0.80. 1=yes, 0=no.
Time Frame: 12 months post randomization
Population: All randomized participants who were taking statins at the time of randomization.
Measure: Number; unit: percent with good adherence
Arm/Group | Usual Care (UC) | Interactive Voice Recognition (IVR) | Enhanced IVR (IVR+)
Number analyzed (Participants) | 5484 | 5453 | 5429
percent with good adherence
  Overall | 32.9 | 35.9 | 35.8
  baseline adherence <=0.40 | 21.5 | 22.6 | 21.8
  baseline adherence 0.4-0.75 | 36.2 | 39.4 | 40.1
  baseline adherence 0.75-0.90 | 58.1 | 63.5 | 62.6
Statistical Analysis 1: Comparison: Usual Care (UC) vs Interactive Voice Recognition (IVR); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.002, Regression, Logistic — Adjusted for site, gender, age, total number of prescription medications patient is taking, comorbid diabetes/CVD, and baseline statin adherence; Odds Ratio (OR) = 1.14, 95% CI 2-sided [1.05 to 1.24] — Adjusted odds ratio for good adherence in IVR group versus UC group, calculated as IVR - UC
Statistical Analysis 2: Comparison: Usual Care (UC) vs Enhanced IVR (IVR+); [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.16, 95% CI 2-sided [1.06 to 1.26] — Adjusted odds ratio for good adherence in IVR+ group versus UC group, calculated as IVR+ - UC

4. Secondary Outcome: Percentage With Good (>80%) ACEI/ARB Adherence
Description: Binary indicator of good ACEI/ARB adherence, defined as an mMPR>0.80. 1=yes, 0=no.
Time Frame: 12 months post randomization
Population: All randomized participants who were taking an ACEI or an ARB at the time of randomization
Measure: Number; unit: Percent with good adherence
Arm/Group | Usual Care (UC) | Interactive Voice Recognition (IVR) | Enhanced IVR (IVR+)
Number analyzed (Participants) | 4330 | 4370 | 4323
Percent with good adherence
  Overall | 37.4 | 40.3 | 41.6
  Baseline adherence <=0.50: number analyzed (Participants) | 2111 | 2123 | 2155
  Baseline adherence <=0.50 | 24.5 | 27.0 | 28.2
  Baseline adherence 0.50-0.75: number analyzed (Participants) | 1049 | 1059 | 1058
  Baseline adherence 0.50-0.75 | 48.4 | 51.1 | 52.0
  Baseline adherence 0.75-0-.90: number analyzed (Participants) | 723 | 680 | 657
  Baseline adherence 0.75-0-.90 | 59.7 | 62.0 | 66.8
Statistical Analysis 1: Comparison: Usual Care (UC) vs Interactive Voice Recognition (IVR); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.014, Regression, Logistic — adjusted for site, gender, age, total number of prescription medications participant was taking, comorbid diabetes/CVD, baseline ACEI/ARB adherence; Odds Ratio (OR) = 1.12, 95% CI 2-sided [1.02 to 1.23] — Adjusted odds ratio for good adherence in IVR group versus UC group, calculated as IVR - UC
Statistical Analysis 2: Comparison: Usual Care (UC) vs Enhanced IVR (IVR+); [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.21, 95% CI 2-sided [1.10 to 1.32] — Adjusted odds ratio for good adherence in IVR group versus UC group, calculated as IVR - UC

5. Secondary Outcome: Systolic Blood Pressure (SBP)
Description: Mean of last 5 SBP measurements captured in the electronic medical record for the 12 months post randomization.
Time Frame: 12-months post randomization
Population: The analysis sample was restricted to ACEI/ARB users with at least one post intervention SBP measurement recorded in the EMR. We did not impute any missing data.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Interactive Voice Recognition (IVR): ACEI/ARB users in IVR arm .
Arm/Group | Usual Care (UC) | Interactive Voice Recognition (IVR) | Enhanced IVR (IVR+)
Number analyzed (Participants) | 3980 | 3980 | 3971
mm Hg
  Overall | 129.2 (13.1) | 128.6 (13.2) | 129.0 (13.2)
  Baseline SBP<=130mmHg: number analyzed (Participants) | 2111 | 2123 | 2155
  Baseline SBP<=130mmHg | 123.5 (10.7) | 122.8 (11.1) | 123.4 (11.1)
  Baseline SBP 130-140mmHg: number analyzed (Participants) | 1049 | 1059 | 1058
  Baseline SBP 130-140mmHg | 132.8 (10.7) | 132.2 (10.1) | 132.7 (10.1)
  Baseline SBP>140mmHg: number analyzed (Participants) | 723 | 680 | 657
  Baseline SBP>140mmHg | 140.6 (13.3) | 140.4 (13.2) | 140.9 (13.2)
Statistical Analysis 1: Comparison: Usual Care (UC) vs Interactive Voice Recognition (IVR); We conducted separate primary analyses of each of IVR and IVR+ versus usual care at the .025 level of significance to assure a trial-wide error rate of .05. This analysis summary is for the IVR versus UC comparison only. Also, we only report results here for the full sample, and not also separately for the 3 baseline SBP level groups; Test type: Superiority or Other; p = .041, Regression, Linear — As noted above, the a priori threshold for statistical significance for this test was .025; Adjusted for site, gender, age, total number of prescription medications patient is taking, comorbid diabetes/CVD, and baseline SBP group; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.0 to 0.0]
Statistical Analysis 2: Comparison: Usual Care (UC) vs Enhanced IVR (IVR+); We conducted separate primary analyses of each of IVR and IVR+ versus usual care at the .025 level of significance to assure a trial-wide error rate of .05. This analysis summary is for the IVR+ versus UC comparison only. Also, we only report results here for the full sample, and not also separately for the 3 baseline SBP level groups; Test type: Superiority or Other; p = .93, Regression, Linear — As noted above, the a priori threshold for statistical significance for this test was .025; Adjusted for site, gender, age, total number of prescription medications participant is taking, comorbid diabetes/CVD, and baseline SBP group; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-.5 to .5]

6. Secondary Outcome: Percentage With Good (<140/90 mmHg) Blood Pressure Control
Description: Using the mean of last 5 available blood pressure measurements post randomization, we defined BP control as a means systolic BP <140 mmHg and a mean diastolic BP < 90 mmHg.
Time Frame: 12 months post randomization
Population: All randomized participants who were taking an ACEI or an ARB at the time of randomization and who had at least one post randomization BP recorded in the EMR. Missing data were not imputed.
Measure: Number; unit: percentage of subjects with good control
Arm/Group | Usual Care (UC) | Interactive Voice Recognition (IVR) | Enhanced IVR (IVR+)
Number analyzed (Participants) | 3980 | 3980 | 3971
percentage of subjects with good control
  Overall | 81.1 | 82.1 | 81.3
  Baseline SBP<=130 mmHg | 93.7 | 94.0 | 92.9
  Baseline SBP 130-140 mmHg | 78.4 | 78.4 | 78.3
  Baseline SBP>140 mmHg | 49.2 | 52.4 | 50.2
Statistical Analysis 1: Comparison: Usual Care (UC) vs Interactive Voice Recognition (IVR); [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = .404, Regression, Logistic — As noted above, the a priori threshold for statistical significance for this test was .025; [statistical method as in outcome 5, analysis 2]; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.93 to 1.19]
Statistical Analysis 2: Comparison: Usual Care (UC) vs Enhanced IVR (IVR+); [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = .54, Regression, Logistic — As noted above, the a priori threshold for statistical significance for this test was .025; [statistical method as in outcome 5, analysis 2]; Odds Ratio (OR) = .96, 95% CI 2-sided [.85 to 1.09]

7. Secondary Outcome: Post Intervention Low Density Lipoprotein (LDL) Level
Description: We used the latest LDL (fasting or nonfasting) available during 12 months post randomization. no missing data were imputed.
Time Frame: 12 months post randomization
Population: All randomized participants who were taking statin at the time of randomization and who had at least one post randomization LDL measurement recorded in the EMR. Missing data were not imputed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Usual Care (UC) | Interactive Voice Recognition (IVR) | Enhanced IVR (IVR+)
Number analyzed (Participants) | 4621 | 4610 | 4545
mg/dL
  Overall | 92.4 (35.3) | 91.8 (34.0) | 91.3 (33.3)
  Baseline LDL <=80 mg/dL: number analyzed (Participants) | 1815 | 1769 | 1734
  Baseline LDL <=80 mg/dL | 75.5 (26.1) | 75.5 (25.7) | 75.6 (26.1)
  Baseline LDL 80-100 mg/dL: number analyzed (Participants) | 1155 | 1224 | 1193
  Baseline LDL 80-100 mg/dL | 92.0 (27.8) | 91.5 (25.9) | 90.7 (24.9)
  Baseline LDL>100 mg/dL: number analyzed (Participants) | 1352 | 1329 | 1346
  Baseline LDL>100 mg/dL | 114.9 (37.9) | 113.0 (37.9) | 111.4 (36.6)
Statistical Analysis 1: Comparison: Usual Care (UC) vs Interactive Voice Recognition (IVR); We conducted separate primary analyses of each of IVR and IVR+ versus usual care at the .025 level of significance to assure a trial-wide error rate of .05. This analysis summary is for the IVR versus UC comparison only. Also, we only report results here for the full sample, and not also separately for the 3 baseline LDL subgroups; Test type: Superiority or Other; p = .38, Regression, Linear — As noted above, the a priori threshold for statistical significance for this test was .025; Adjusted for site, gender, age, total number of prescription medications participant is taking, comorbid diabetes/CVD, and baseline LDL group; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.8 to 0.7]
Statistical Analysis 2: Comparison: Usual Care (UC) vs Enhanced IVR (IVR+); We conducted separate primary analyses of each of IVR and IVR+ versus usual care at the .025 level of significance to assure a trial-wide error rate of .05. This analysis summary is for the IVR+ versus UC comparison only. Also, we only report results here for the full sample, and not also separately for the 3 baseline LDL level subgroups; Test type: Superiority or Other; p = .019, Regression, Linear — As noted above, the a priori threshold for statistical significance for this test was .025; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-2.7 to -0.2] — MeanLDL levels were sig lower for IVR+ participants than for UC participants. In subgroup analyses this difference was most pronounced in those individuals with baseline LDL levels above 100 mg/dL (adj diff=-3.6 mg/dL, 95%CI= (-5.9, -1.3), p=.002)

8. Secondary Outcome: Percentage With Good (<=100mg/dL) Low Density Lipoprotein (LDL) Control
Description: Using the last LDL measurement (fasting or nonfasting) available in the EMR post randomization, we defined good control as an LDL level <= 100 mg/dL.
Time Frame: 12 months post randomization
Population: All randomized participants who were taking a statin at the time of randomization and who had at least one post randomization LDL measurement recorded in the EMR. Missing data were not imputed.
Measure: Number; unit: percentage with controlled LDL
Arm/Group | Usual Care (UC) | Interactive Voice Recognition (IVR) | Enhanced IVR (IVR+)
Number analyzed (Participants) | 4621 | 4610 | 4545
percentage with controlled LDL
  Overall | 69.1 | 69.8 | 70.4
  Baseline LDL <=80 mg/dL | 88.4 | 88.0 | 88.1
  Baseline LDL 80-100 mg/dL | 73.7 | 74.0 | 74.9
  Baseline LDL > 100 mg/dL | 39.9 | 43.5 | 44.1
Statistical Analysis 1: Comparison: Usual Care (UC) vs Interactive Voice Recognition (IVR); We conducted separate primary analyses of each of IVR and IVR+ versus usual care at the .025 level of significance to assure a trial-wide error rate of .05. This analysis summary is for the IVR versus UC comparison only. Also, we only report results here for the full sample, and not also separately for the 3 baseline LDL level subgroups; Test type: Superiority or Other; p = .59, Regression, Logistic — As noted above, the a priori threshold for statistical significance for this test was .025; [statistical method as in outcome 7, analysis 1]; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.93 to 1.13]
Statistical Analysis 2: Comparison: Usual Care (UC) vs Enhanced IVR (IVR+); [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = .058, Regression, Logistic — As noted above, the a priori threshold for statistical significance for this test was .025; [statistical method as in outcome 7, analysis 1]; Odds Ratio (OR) = 1.10, 95% CI 2-sided [1.00 to 1.22] — Though higher for the IVR+ group, LDL control did not differ significantly between the IVR+ and UC arms. Among those with poor initial control, however, control was sig better for the IVR+ arm (OR = 1.21, 95%CI = (1.04, 1.42), p=.015)

ADVERSE EVENTS:
Time Frame: 12 months post randomization
Groups:
- Usual Care (UC): usual medical care
- Interactive Voice Recognition (IVR): usual care plus automated phone calls
- Enhanced IVR (IVR+): usual care plus automated phone calls plus educational mailings and mail follow-up for persistent nonadherence
Arm/Group | Usual Care (UC) | Interactive Voice Recognition (IVR) | Enhanced IVR (IVR+)
All-Cause Mortality (participants affected / at risk) | 141/7255 | 146/7247 | 140/7250
Serious Adverse Events (participants affected / at risk) | 25/7255 | 21/7247 | 22/7250
Other Adverse Events (participants affected / at risk) | 0/7255 | 0/7247 | 0/7250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Usual Care (UC) (N=7255) | Interactive Voice Recognition (IVR) (N=7247) | Enhanced IVR (IVR+) (N=7250)
potential ACEI/ARB related hospitalization (Vascular disorders) | 24/4330 (24) | 19/4370 (19) | 20/4323 (20) — organ system categorization is incomplete. this includes hospitalization for acute renal failure, angioedema, anaphylactic shock, and anaphylactic hypotension
potential statin related hospitalization (Hepatobiliary disorders) | 1/3980 (1) | 2/3980 (2) | 2/3971 (2) — specifically includes hospitalizations for liver failure or cirrhosis rhabdomyolysis as a primary discharge diagnosis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No